CLINICAL TRIAL: NCT04735666
Title: European TauroPace Registry - University of Schleswig-Holstein Prospective Observational Clinical Study
Acronym: ETPR
Status: Recruiting | Type: Observational
Sponsor: University of Kiel (Other)
Collaborators: University of Luebeck (Other)
Responsible Party: Principal Investigator, Prof. Dr. Hendrik Bonnemeier, Coordinating Investigator ETPR, University of Kiel
Other Study IDs: 1.1
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: CIED Related Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: TauroPace™ — TauroPace™ is intended to be used as a disinfecting solution during any CIED related surgery procedure or handling of any uncoated or silicon-, epoxy- or polyurethane-coated CIED (including its components, e.g., leads) made of titan or stainless steel in any adult patient requiring or carrying a CIED.

SUMMARY:
University of Schleswig-Holstein Campus Kiel is sponsoring the European TauroPace Registry. This investigator-initiated local, prospective, non-interventional, multi-center study includes patients undergoing cardiac implantable electronic placement including and not limited to placement, revision with the aim to upgrade or downgrade, generator substitution, additional lead placement, revision or extraction (procedure) with adjunct TauroPace. It is planned to include a total of at least 2300 procedures (valid for safety analysis).

DETAILED DESCRIPTION:
This study is performed as an all-case investigation. The treatment is performed based on the SOPs (Appendix Study Protocol). The standard observation period is 3 months from the 1st treatment. Safety and effectiveness are evaluated at 3rd and 12th month. In addition, the extension observation is carried out once a year for 3 years at the longest to collect information on safety and effectiveness as long as CIED treatment continues. When the treatment ends (extraction of all hardware), observation of a patient ends. For each patient, the investigator records data as defined in the protocol at each evaluation point by using a unique Case Report Form (CRF) system. The duration of the study is estimated at 10 years (registry).

ELIGIBILITY:
Inclusion Criteria:

* Use of TauroPace™ is indicated and not contra-indicated according to its current Instructions For Use (IFU)
* Participant is eligible for a CIED related surgery procedure.

Exclusion Criteria:

* Age<18years
* Participant incapable of signing Patient Informed Consent (mentally or physically) or does not sign.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consist of every subsequent participant eligible for any CIED related surgery with TauroPace™
Sampling Method: Non-Probability Sample
Enrollment: 2300 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2030-01-30 (Estimated); Study Completion 2030-01-30 (Estimated)

PRIMARY OUTCOMES:
CIED infections | three months
  CIED infections occurring in an observation period of three months after any CIED related surgical procedure in different CIED using a regimen with surface disinfection of CIEDs and irrigation of the surgical site (pocket) with a taurolidine containing antimicrobial compound adjunct.

SECONDARY OUTCOMES:
CIED infections | 12 months
  CIED infections occurring in an observation period of 12 months after any CIED related surgical procedure in different CIED using a regimen with surface disinfection of CIEDs and irrigation of the surgical site (pocket) with a taurolidine containing antimicrobial compound adjunct.
CIED infections | 36 months
  CIED infections occurring in an observation period of 36 months after any CIED related surgical procedure in different CIED using a regimen with surface disinfection of CIEDs and irrigation of the surgical site (pocket) with a taurolidine containing antimicrobial compound adjunct.
AE | 3, 12 and 36 months
  Adverse events (complications) during 3, 12 and 36 months follow-up
All-cause mortality | 3, 12 and 36 months
  Allcause mortality during 3, 12 and 36 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik Bonnemeier, PhD, Principal Investigator — University of Kiel - Medical Faculty
Locations (8):
- Landeskrankenhaus Wiener Neustadt, Wiener Neustadt, Austria
- Louis Pradel Hospital, Lyon, Bron, France
- Germany (4):
  - Krankenhaus Landshut Achdorf, Landshut, Bavaria
  - Helios Klinik Cuxhaven, Cuxhaven, Lower Saxony
  - Helios Klinik Wesermarsch, Nordenham, Lower Saxony
  - University Hospital Schleswig-Holstein, Kiel, Schleswig-Holstein
- Ospedale Regionale San Maurizio, Bolzano, Trentino-Alto Adige, Italy
- Great Western Hospitals NHS Foundation Trust, Swindon, United Kingdom

IPD SHARING:
Plan to Share IPD: No
participant data is recorded in a pseudonymous manner in the centre, before statistical analysis data is anonymized

REFERENCES:
- [Derived] Vonthein R, Baldauf B, Borov S, Lau EW, Giaccardi M, Assadian O, Haddad C, Chevalier P, Bode K, Foley P, Thomas H, Campbell NG, Fichtner S, Donazzan L, Pescoller F, Oberhollenzer R, Cemin R, Bonnemeier H. Taurolidine-containing solution for reducing cardiac implantable electronic device infection-early report from the European TauroPace registry. J Cardiothorac Surg. 2024 Oct 4;19(1):592. doi: 10.1186/s13019-024-03059-1. PMID 39367427
- See also: domain of the EuropeanTauroPace Registry — http://www.etpr.eu